CLINICAL TRIAL: NCT04450459
Title: Impact of Ergospirometric Oxygen Uptake Under Exercise as Diagnostic Marker of Cardiac Ischemia in Patients With Stable Angina Compared to Non Invasive and Invasive (FFR) Measurement of Ischemia
Brief Title: Impact of Spiroergometer Parameters as Diagnostic Marker of Cardiac Ischemia in Pts. With Stable Angina Compared to FFR.
Acronym: ADVANCE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Jena University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: SMW 08
Record Dates: First submitted 2020-06-25; First posted 2020-06-29 (Actual); Last update posted 2022-08-11 (Actual); Status verified 2022-08

CONDITIONS: Stable Angina
Keywords: FFR Measurement; exercise testing, ergospirometer
MeSH Terms: conditions — Angina, Stable

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — EDTA Blood, Serum,

INTERVENTIONS:
Diagnostic Test: ergospirometer test — ergospirometric test will be done before cardiac catheterisation and invasive measurement of FFR

SUMMARY:
In Patients with stable Angina pectoris CCS 1-3 exercise testing for ischemia detection is widely used despite the known limitations. Measurement of the FFR is invasive but gold standard for Ischemia detection.

Adding of parameters of spiroergometer might help to improve diagnostic accuracy of non invasive exercise testing. Therefore the trial is evaluating diagnostic accuracy of spiroergometric parameters compared to invasive FFR measurement.

ELIGIBILITY:
Inclusion Criteria:

* stable Angina (CCS >1-3) with suspected CAD or
* dyspnoea at exertion NYHA >2 or
* signs of ischemia within SPECT or exercise electrocardiography
* willingness to participate in the trial

Exclusion Criteria:

* Unstable angina or myocardial infarction within the last 2 weeks
* inability to perform bicycle exercise test
* significant valvular disease
* HOCM
* av- block >I degree
* asthma bronchiales

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: patients with suspected CAD presenting for diagnostic testing/ coronary angiography
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2019-01-02 (Actual); Primary Completion 2023-01 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
double slope sign of ΔV̇O2/ΔWR-Increase | baseline
  double slope sign of ΔV̇O2/ΔWR by ergospirometer test

CONTACTS AND LOCATIONS:
Overall Officials: Sven Möbius-Winkler, MD, Principal Investigator — Universityhospital Jena
Locations (1):
- Universityhospital, Jena, Germany

IPD SHARING:
Plan to Share IPD: No